CLINICAL TRIAL: NCT02048540
Title: Phase 2 Study of Neoadjuvant Bevacizumab Plus DOF Versus DOF in Local Advanced Gastric Carcinoma and Its Association With Circulating Tumor Cell
Brief Title: Neoadjuvant Bev Plus DOF vs DOF in LAGC and Its Association With Circulating Tumor Cell
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, DuNan, professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC neoadjuvant bev CTC; BSC2013-dunan (Other: Beijing science commission)
Record Dates: First submitted 2014-01-25; First posted 2014-01-29 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Locally Advanced Gastric Carcinoma
MeSH Terms: interventions — Bevacizumab; Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- bevacizumab plus DOF (Experimental): patients receive bev +DOF pre and post surgery up to total 6 cycles
  Interventions: Biological: Bevacizumab; Drug: docetaxel oxaliplatin 5-FU CF; Procedure: Gastrectomy
- DOF (Active Comparator): patients receive DOF pre and post surgery up to total 6 cycles
  Interventions: Drug: docetaxel oxaliplatin 5-FU CF; Procedure: Gastrectomy

INTERVENTIONS:
Biological: Bevacizumab — Bev (5 mg/kg, d1) every 3 weeks, up to 2-4 cycles preoperation, and another 2-4 cycles postoperation up to total 6 cycles.
  Arms: bevacizumab plus DOF
Drug: docetaxel oxaliplatin 5-FU CF — docetaxel, 75 mg/m2, iv, d1; oxaliplatin, 85 mg/m2, iv, d1; 5-FU, iv infusion 600 mg/m2 and iv injection 400mg/m2, d1-2; CF, 200 mg/m2, d1 and d2 each 3-week, up to 2-4 cycles preoperation, and another 2-4 cycles postoperation up to total 6 cycles.
Procedure: Gastrectomy

SUMMARY:
Background Local advanced gastric carcinoma (LAGC) is suggested to be potentially cured by R0 resection, and neoadjuvant chemotherapy can increase the R0 resection rate but not enough. Bevacizumab (Bev), an anti-tumor angiogenesis monoclonal antibody, combined with chemotherapy has been shown effective in advanced GC. In addition, CTC has been suggested as an indicator of the anti-tumor drugs' efficacy. Therefore, in this study, the investigators plan to evaluate the efficacy and safety of neoadjuvant Bev plus docetaxel/oxaliplatin/5-FU/CF (DOF) versus DOF in mainly gastric antrum LAGC, and to investigate whether CTC is an effectiveness indicator.

Methods 86 patients diagnosed as IIIb-IIIc GC have been enrolled and randomly assigned (1:1) to receive neoadjuvant Bev (5 mg/kg, d1) plus DOF (docetaxel, 75 mg/m2, iv, d1; oxaliplatin, 85 mg/m2, iv, d1; 5-FU, iv infusion 600 mg/m2 and iv injection 400mg/m2, d1-2; CF, 200 mg/m2, d1 and d2) or DOF each 3-week, up to 2-4 cycles preoperation, and another 2-4 cycles postoperation up to total 6 cycles. The primary endpoint is R0 resection rate. CTC was detected every 8 weeks. All patients signed the informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced adenocarcinoma of the stomach.
* Age of 18 to 70, Karnofsky score higher than 80.
* T3-4，N1-3，M0 (AJCC 7th), potentially resectable.
* No severe functional damage of major organ, normal blood cell, normal liver and kidney function.

Exclusion Criteria:

* Clinical findings of distant metastasis or Peritoneal carcinomatosis
* Prior systemic (chemo- or targeted) treatment. Prior radiotherapy to the upper abdomen
* Previous malignancy within 5 years, with the exception of adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer
* Upper gastrointestinal bleeding
* Any contraindication to treatment with docetaxel, 5-fu or oxaliplatin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
R0 resection rate | 6-12 weeks after administration

SECONDARY OUTCOMES:
pCR rate | Day 1 after surgery
OS | 3 years after surgery
DFS | 3 years after surgery
ORR | 6 weeks after administration
safety of peroperative treatment and surgery | from first administration to 28 days after last administration

OTHER OUTCOMES:
circulating tumor cell number change | 6 weeks
  to investigate the circulating tumor cell number change before and after neoadjuvant therapy and whether it's an effectiveness and survival predictor in LAGC

CONTACTS AND LOCATIONS:
Overall Officials: Nan Du, Phd, Principal Investigator — First Affiliated Hospital, Chinese PLA General Hospital
Locations (1):
- First Affiliated Hospital, Chinese PLA General Hospital, Beijing, Beijing Municipality, China